CLINICAL TRIAL: NCT03362801
Title: SArcopenia, Mobility, PHYsical Activity and Post-operative Risk of Bladder Carcinoma in the Elderly
Acronym: SAMPHYR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SAMPHYR 16-181.
Record Dates: First submitted 2017-03-07; First posted 2017-12-05 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2023-09

CONDITIONS: Sarcopenia; Bladder Cancer
Keywords: physical activity; elderly
MeSH Terms: conditions — Sarcopenia; Urinary Bladder Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sarcopenic (Other): sarcopenic status the day before cystectomy.
  Interventions: Diagnostic Test: sarcopenia and mobility measurement
- not sarcopenic (Other): sarcopenic status the day before cystectomy.
  Interventions: Diagnostic Test: sarcopenia and mobility measurement

INTERVENTIONS:
Diagnostic Test: sarcopenia and mobility measurement — walking speed, grip strength and BIA. QAPPA questionnaire (validated in French in the elderly) and the objective measurement of the time of activity and rest on a week per wrist actimeter.
  Comprehensive Geriatric Assessment

SUMMARY:
Sarcopenia is associated with lower prognosis in solid tumors, but this has not been studied in bladder carcinoma requiring cystectomy.

According to EWGSOP recommendations, the diagnosis of sarcopenia is based on walking speed, grip strength and muscle mass. These three elements can easily be measured (specially muscle mass measurement by bioimpedencemetry or tomodensitometry).

This cohort study will collect clinical complementary elements to better understand the associated factors present with sarcopenia, in order to prepare an interventional preoperative physical reconditioning study.

The mobility measurement will be carried out by the QAPPA questionnaire (validated in French in the elderly) and the quantitative measurement of activity and rest hours during a week by a wrist actimeter.

Standardized geriatric data will also be collected: ADL, IADL for autonomy, MMSE for cognitive status, nutritional status (% weight loss, BMI), pain, GDS15 for depression screening, updated Charlson Comorbidity Index to identify polypathology and The STOPP tool for potentially inappropriate medication.

Post-operative morbidity mortality at 30 days will be evaluated according to Clavien-Dindo classification. Investigators will also evaluate 6 months geriatric complications : falls, loss of autonomy and decreased mobility and physical activity, cognitive degradation, undernutrition, institutionalization

ELIGIBILITY:
Inclusion Criteria:

* confirmed urothelial bladder carcinoma ( RTUV)

  * indication of radical cystectomy
  * Able, informed and with informed consent for the study
  * affiliated to the social security system
  * talking French

Exclusion Criteria:

* Life expectancy <6 months

  * other active malignant tumors or other severe concomitant chronic pathologies affecting the general condition of the patient and / or likely to limit compliance with the requirements of the study.
  * treatments incompatible with the study: previous corticosteroid treatment prolonged for more than one month (induces iatrogenic sarcopenia).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
post-operative morbidity | at 30 days
  evaluated according to Clavien-Dindo classification
post-operative mortality | at 30 days

SECONDARY OUTCOMES:
post-operative complications | 8 months
  Impact of dependancy (PS / ADL / IADL)
post-operative complications | 8 months
  physical activity scores (QAPPA) Questionnaire d'activité physique pour les personnes âgées in French validated in French population - total score is used
post-operative complications | 8 months
  physical performance (PBP)
post-operative complications | 8 months
  fatigue (BFI) Brief Fatigue Inventory questionnaire
post-operative complications | 8 months
  history of fall
post-operative complications | 8 months
  pain (visual analogic scale for pain 0 to 10)
post-operative complications | 8 months
  hours of mobility (actimetry)
post-operative complications | 8 months
  hours of daily rest (actimetry) measured during 3 consecutives days
post-operative complications | 8 months
  Actimetry
post-operative complications | 8 months
  nutritional status (nutritional grade 2 or 4 according to SFNEP Société Francophone Nutrition Clinique et Métabolisme )
post-operative complications | 8 months
  cognitive status (normal or not)
post-operative complications | 8 months
  polymedication (≥5 / day)
post-operative complications | 8 months
  comorbidities (updated charlson)
post-operative complications | 8 months
  inappropriate prescriptions (STOPP)
impedancemetric value | 2 months
  Concordance of values (attribution of sarcopenic / non-sarcopenic groups) with impedancemetric value
sarcopenic status | between baseline; preoperative and at 6 months post-operative
  evolution of sarcopenic status
quality of life scores | preoperative and 6-month post-operative
  EORTC QLQ-ELD14 (assessment of health-related quality of life elderly patients with cancer with 14 items)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Caen University Hospital, Caen
  - APHM, Marseille
  - Rouen UH, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Audisio RA, Bozzetti F, Gennari R, Jaklitsch MT, Koperna T, Longo WE, Wiggers T, Zbar AP. The surgical management of elderly cancer patients; recommendations of the SIOG surgical task force. Eur J Cancer. 2004 May;40(7):926-38. doi: 10.1016/j.ejca.2004.01.016. PMID 15093567
- [Result] Huisman MG, van Leeuwen BL, Ugolini G, Montroni I, Spiliotis J, Stabilini C, de'Liguori Carino N, Farinella E, de Bock GH, Audisio RA. "Timed Up & Go": a screening tool for predicting 30-day morbidity in onco-geriatric surgical patients? A multicenter cohort study. PLoS One. 2014 Jan 24;9(1):e86863. doi: 10.1371/journal.pone.0086863. eCollection 2014. PMID 24475186
- [Result] Shachar SS, Williams GR, Muss HB, Nishijima TF. Prognostic value of sarcopenia in adults with solid tumours: A meta-analysis and systematic review. Eur J Cancer. 2016 Apr;57:58-67. doi: 10.1016/j.ejca.2015.12.030. Epub 2016 Feb 13. PMID 26882087
- [Result] Psutka SP, Carrasco A, Schmit GD, Moynagh MR, Boorjian SA, Frank I, Stewart SB, Thapa P, Tarrell RF, Cheville JC, Tollefson MK. Sarcopenia in patients with bladder cancer undergoing radical cystectomy: impact on cancer-specific and all-cause mortality. Cancer. 2014 Sep 15;120(18):2910-8. doi: 10.1002/cncr.28798. Epub 2014 May 19. PMID 24840856
- [Result] Smith AB, Deal AM, Yu H, Boyd B, Matthews J, Wallen EM, Pruthi RS, Woods ME, Muss H, Nielsen ME. Sarcopenia as a predictor of complications and survival following radical cystectomy. J Urol. 2014 Jun;191(6):1714-20. doi: 10.1016/j.juro.2013.12.047. Epub 2014 Jan 11. PMID 24423437